CLINICAL TRIAL: NCT01893944
Title: Applicability of Video Games and Vibrational Therapy in Reducing Pain Secondary to Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 07694812.7.0000.5501
Record Dates: First submitted 2013-06-24; First posted 2013-07-09 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pain
Keywords: Breast cancer; vibratory therapy; virtual reality
MeSH Terms: conditions — Pain; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Virtual Reality (Experimental): - Participate in this group 20 women to be treated by means of games Xbox 360 ®, attributed to this, custom applications using virtual and augmented reality to be developed.
  Interventions: Other: virtual reality
- Vibration therapy (Experimental): - participate in this group 20 women who will undergo 15 minutes of continuous vibration by vibration of the upper mantle, with a frequency of 40 Hz, 3 function and intensity tolerable, keeping the limb supported and raised to 120 °.
  Interventions: Other: virtual reality
- control group (Active Comparator): - participate in this group 20 women who are treated with conventional cinesioterapia through muscle stretching exercises, dissociation girdle, active and active-assisted exercises for groups flexors, extensors, abductors and adductors of the upper limbs, which will be three series 10 repetitions for each exercise.
  Interventions: Other: virtual reality

INTERVENTIONS:
Other: virtual reality — customized applications using virtual and augmented reality to be developed.

SUMMARY:
To evaluate the influence of virtual reality and vibrational therapy in reducing pain intensity secondary to breast cancer before and after application of treatment protocols, through biomedical instrumentation.

DETAILED DESCRIPTION:
After physiotherapy assessment individuals will be randomly divided into three groups: Group Virtual Reality - Cinesioterapia (G1), Group Vibration Therapy - Cinesioterapia (G2) and Control Group (G3), which will be submitted to the respective treatment protocols. Group Virtual Reality Cinesioterapia (G1) participate in this group 20 women will be treated through the games Xbox 360 ®, attributed to this, customized applications using virtual and augmented reality to be developed. Vibration Therapy Group - Cinesioterapia (G2) - will participate in this group 20 women who will undergo 15 minutes of continuous vibration through the blanket vibrating members higher, with frequency 40 Hz, 3 function and intensity tolerable, keeping the limb supported and elevated to 120 º. At the end held muscle stretching exercises, dissociation of shoulder girdle and upper limb exercises assets. Control group (G3) - participate in this group 20 women who are treated with conventional cinesioterapia through muscle stretching exercises for flexors, extensors, adductors and abductors shoulder for 20 seconds each; dissociation girdle; financial assets and Active assisted for groups flexors, extensors, abductors and adductors of the upper limbs, which will be performed three sets of 10 repetitions for each exercise. Implementation of treatment protocols for the groups G1, G2 and G3 will run for two weeks, being Monday through Friday feira.totalizando 10 consecutive treatment sessions lasting 30 minutes each session. You will be prompted to patients groups G1, G2 and G3 to respond individually and without any aid the visual numeric scale of pain, 10 minutes pre-therapy, 15 minutes after the start and 10 minutes after the end of therapy. Patients will undergo the assessment of pain, electromyographic activity of muscles, muscle strength, range of motion analysis and perimetry in the first day of treatment, and after completing all the sessions patients were reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent surgery for unilateral mastectomy and axillary lymphadenectomy modified in a period exceeding one year;
* Submit medical referral;
* Which are not performing radiotherapy or chemotherapy;
* Age 40-70 years;
* Reporting pain, intermittent, prolonged duration and intensity that limits the ADL;
* Lymphedema in the ipsilateral upper limb surgery;
* To agree and sign the Statement of Consent

Exclusion Criteria:

* Individuals who fail to provide medical referral;
* Be a carrier of other types of cancer;
* Have undergone other types of surgery removal of breast cancer; - be doing chemotherapy or radiotherapy;
* Do not complain of pain symptoms and lymphedema;
* Presenting severe joint lock.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain secondary to breast cancer | one year
  Expect positive results of this research on the reduction of pain as well as physical and functional complications caused by surgery for breast cancer, enabling a better quality of life for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Lersm, Ip&D, São José dos Campos, São Paulo, Brazil